CLINICAL TRIAL: NCT06497647
Title: Outcome of Treatment of Monosymptomatic Nocturnal Enuresis in Children Using Imipramine Alone Versus Sulbutiamine Alone Versus Imipramine Plus Sulbutiamine : Prospective Comparative Study
Brief Title: New Treatment for Nocturnal Enuresis in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Loai Mohammed Abd Al-Hamied, resident of urology , sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med-24-06-05MS
Record Dates: First submitted 2024-07-01; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Nocturnal Enuresis in Children
Keywords: treatment of monosymptomatic nocturnal enuresis in children using sulbutiamine
MeSH Terms: interventions — sulbutiamine; Imipramine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): this group will receive imipramine alone
  Interventions: Drug: Imipramine
- group B (Active Comparator): this group will receive sulbutiamine alone
  Interventions: Drug: Sulbutiamine
- group C (Active Comparator): this group will receive sulbutiamine plus imipramine
  Interventions: Drug: Sulbutiamine; Drug: Imipramine

INTERVENTIONS:
Drug: Sulbutiamine — sulbutiamine will be used by oral route 100 mg daily for 1 month and follow up will be done every 1 month till 3 months.
  it will be used alone in group B and combined with imipramine in group C
  Arms: group B; group C
Drug: Imipramine — imipramine will be used by oral route 25 mg daily for 1 month and follow up will be done every 1 month till 3 months.
  it will be used alone in group A and combined with sulbutiamine in group C
  Arms: group A; group C

SUMMARY:
The aim of the study is to evaluate the role of sulbutiamine in treatment of monosymptomatic nocturnal enuresis in children by using it alone or as a combination therapy with tricyclic antidepressants (imipramine+sulbutiamine).

ELIGIBILITY:
Inclusion Criteria:

* Age : 6 - 18 years old.
* All children diagnosed by Primary monosymptomatic nocturnal enuresis in this age group.

Exclusion Criteria:

* Secondary nocturnal enuresis (child who has been continent for at least 6 months before the onset of bedwetting ).
* congenital anomalies (Posterior urethral valve , ectopic ureter , ectopia vesica ,…)
* history of previous lower urinary tract surgery (Multiple hypospadias surgeries ,…, )
* neurogenic bladder (as underactive bladder ).and urge incontinence.
* presence of post-void residual urine greater than 20% of functional bladder capacity.
* history or evidence of disorders in other organs such as (cardiovascular system disease), liver , psychological problems , evident allergic reaction to both medication.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
reduction in the number of wet nights . | the number of wet nights will be measured and compared at the end of each month for 3 months using a calendar fulfilled by the child and his parents.
  A questionnaire which measure the Response to treatment which will be evaluated by the standardization committee of International clildren's continence society (ICCS) as follows :
  * Complete response : 100% reduction
  * Partial response : 50% - 99% reduction
  * Unresponsiveness : 0 - 49% reduction in nocturnal enuresis episodes.
  this will be measured by a questionnaire that will be written according a calendar fulfilled by the child and his parents with comparison of the number of wet nights each month.

SECONDARY OUTCOMES:
determine any side effects of the drugs used in the study | this will be discussed in the follow up that will be done in each month in the outpatient clinic for 3 months.
  asking the child and his parents about any abnormal findings or symptoms appear in the period of the treatment this will be done by a questionnaire that will be fulfilled by the child and his parents.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Faculty of Medecine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided